CLINICAL TRIAL: NCT00451555
Title: A Randomized, Double-Blind, Phase II Trial of Fulvestrant Plus Enzastaurin Versus Fulvestrant Plus Placebo in Aromatase Inhibitor-Resistant Metastatic Breast Cancer
Brief Title: Enzastaurin Plus Fulvestrant vs. Placebo Plus Fulvestrant in Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 10736; H6Q-MC-S023 (Other: Eli Lilly and Company)
Record Dates: First submitted 2007-03-21; First posted 2007-03-23 (Estimated); Results first posted 2019-11-01 (Actual); Last update posted 2019-11-01 (Actual); Status verified 2018-11-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — enzastaurin; Fulvestrant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Enzastaurin + Fulvestrant (Experimental): Participants received Enzastaurin loading dose of 1125 mg, on Day 1 of Cycle 1 only then received Enzastaurin 500 mg orally (QD) once daily in a 28-day cycle.
  Participants received enzastaurin loading dose of 1125 mg, on Day 1 of Cycle 1 only then received Enzastaurin 250 mg orally (BID) twice daily in a 28-day cycle.
  Fulvestrant was given intramuscularly at a loading dose of 500 mg on Day 1 and 250 mg on Day 15 in Cycle 1. Subsequent doses of Fulvestrant 250 mg were given on Day 1 of Cycle 2 and every 28 days thereafter.
  Interventions: Drug: enzastaurin; Drug: fulvestrant
- Fulvestrant + Placebo (Placebo Comparator): Participants received fulvestrant: 500 mg, IM, day 1, 1250 mg, IM, day 15 cycle 1 then 250 mg, IM, every 28 days, until disease progression. Then, participants received placebo, oral, daily.
  Interventions: Drug: placebo; Drug: fulvestrant

INTERVENTIONS:
Drug: enzastaurin — 1125 milligram (mg) loading dose then 250 mg, oral, twice daily (for a total of 500 mg), until disease progression
  Other Names: LY317615
  Arms: Enzastaurin + Fulvestrant
Drug: placebo — oral, daily
  Arms: Fulvestrant + Placebo
Drug: fulvestrant — 500 mg, intramuscular (IM), day 1, 1250 mg, IM, day 15 cycle 1 then 250 mg, IM, every 28 days, until disease progression

SUMMARY:
The primary purpose of this study is to help answer the following research question: whether enzastaurin given together with fulvestrant can help participants who have breast cancer and make the tumor smaller or disappear and for how long.

ELIGIBILITY:
Inclusion Criteria:

* Female participants with a histological-documented diagnosis of locally advanced or metastatic breast cancer. The primary or metastatic tumor must be estrogen response (ER) and/or parathyroid hormone receptor (PtR) positive.

Note: Hormone receptor positivity is defined as ER or PtR greater than 10 fmol/mg by biochemical assay or 10% positive cells by immunohistochemistry

* Participants are resistant to aromatase inhibitors (AI) therapy
* Females with postmenopausal status
* Previous radiation therapy is allowed, but should have been limited
* Measurable or non-measurable disease
* Have a performance status of 0, 1, or 2 on the Eastern Cooperative Oncology Group (ECOG) scale
* Have adequate organ function
* Have an estimated life expectancy of at least 24 weeks
* Must sign an informed consent document

Exclusion Criteria:

* Have had prior treatment with fulvestrant or enzastaurin
* Are receiving concurrent administration of any other antitumor therapy, with the exception of gonadotropin-releasing hormone (GnRH) antagonists.
* Have received treatment within the last 4 weeks with a drug that has not received regulatory approval for any indication at the time of study entry
* Have received supplemental estrogen or progesterone within 4 weeks prior to study entry
* Are hormone estrogen receptor (HER2)-positive
* Are unable to discontinue use of anticoagulants
* Have hypercalcemia
* Have a second primary malignancy that is clinically detectable at the time of consideration for study enrollment
* Have documented central nervous system (CNS) metastases, symptomatic pulmonary lymphangitis, or involvement of more than 1/3 of the liver
* Have a serious concomitant systemic disorder
* Have a serious cardiac condition
* Are unwilling or unable to discontinue use of carbamazepine, phenobarbital, or phenytoin at least 14 days prior to study therapy
* Are unable to swallow tablets.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2007-04-11 (Actual); Primary Completion 2010-12-28 (Actual); Study Completion 2018-10-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (21):
- France (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Besançon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Paris
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint-Herblain
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toulouse
- Germany (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bielefeld
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dresden
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gütersloh
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kiel
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mannheim
- Italy (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Meldola
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Milan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Modena
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rome
- Netherlands (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Amsterdam
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Groningen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Maastricht
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., The Hague
- Spain (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barcelona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lleida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madrid
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Valencia

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- See also: Lilly Clinical Trial Registry — https://vivli.org

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Completers include participants who had died from any cause, who discontinued due to progressive disease or were alive and on study but no longer receiving treatment at end of the study.
Groups:
- Enzastaurin + Fulvestrant: (Initial Therapy) Participants received Enzastaurin loading dose of 1125 mg, on Day 1 of Cycle 1 only then received Enzastaurin 500 mg orally (QD) once daily in a 28-day cycle.
  (Amended Therapy) Participants received enzastaurin loading dose of 1125 mg, on Day 1 of Cycle 1 only then received Enzastaurin 250 mg orally (BID) twice daily in a 28-day cycle.
  Enzastaurin Once Daily Dosing: Participants received Enzastaurin 500 mg QD. Enzastaurin Twice Daily Dosing: Participants received Enzastaurin 500 mg BID. Fulvestrant was given intramuscularly at a loading dose of 500 mg on Day 1 and 250 mg on Day 15 in Cycle 1. Subsequent doses of Fulvestrant 250 mg were given on Day 1 of Cycle 2 and every 28 days thereafter.
- Fulvestrant + Placebo: Participants received fulvestrant: 500 mg, intramuscular (IM), day 1, 1250 mg, IM, day 15 cycle 1 then 250 mg, IM, every 28 days, until disease progression. Then, participants received placebo, oral, daily.
Period: Overall Study
Arm/Group | Enzastaurin + Fulvestrant | Fulvestrant + Placebo
Started | 96 | 60
Received at Least One Dose of Study Drug | 94 | 58
Enzastaurin Twice Daily Dosing (BID) | 39 | 0
Enzastaurin Once Daily Dosing (QD) | 55 | 0
Progressive Disease | 75 | 54
Death | 2 | 0
Completed | 83 | 56
Not Completed | 13 | 4
Not completed — Protocol Violation | 2 | 2
Not completed — Adverse Event | 3 | 1
Not completed — Withdrawal by Subject | 6 | 0
Not completed — Physician Decision | 2 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least one dose of study drug.
Groups:
- Enzastaurin + Fulvestrant BID: Participants received Enzastaurin 1125 mg loading dose then 250 mg, oral, twice daily (BID) (for a total of 500 mg), until disease progression
  Fulvestrant was given intramuscularly at a loading dose of 500 mg on Day 1 and 250 mg on Day 15 in Cycle 1. Subsequent doses of Fulvestrant 250 mg were given on Day 1 of Cycle 2 and every 28 days thereafter.
- Enzastaurin + Fulvestrant QD: Participants received Enzastaurin 1125 mg loading dose then received Enzastaurin once daily (QD) regimen of enzastaurin 500 mg orally QD in a 28-day cycle until disease progression.
  Fulvestrant was given intramuscularly at a loading dose of 500 mg on Day 1 and 250 mg on Day 15 in Cycle 1. Subsequent doses of Ful 250 mg were given on Day 1 of Cycle 2 and every 28 days thereafter.
- Placebo + Fulvestrant BID: Participants received fulvestrant: 500 mg, IM, day 1, 1250 mg, IM, day 15 cycle 1 then 250 mg, IM, every 28 days, until disease progression.
  Then, participants received placebo, oral, daily.
- Total: Total of all reporting groups
Arm/Group | Enzastaurin + Fulvestrant BID | Enzastaurin + Fulvestrant QD | Placebo + Fulvestrant BID | Total
Number analyzed (Participants) | 39 | 55 | 58 | 152
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.2 (9.1) | 66.5 (10.3) | 65.4 (10.0) | 64.9 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 55 | 58 | 152
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 57 | 57
  Not Hispanic or Latino | 39 | 55 | 1 | 95
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1
  White | 38 | 55 | 58 | 151
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Netherlands | 9 | 5 | 6 | 20
  Italy | 7 | 6 | 5 | 18
  France | 11 | 24 | 25 | 60
  Germany | 3 | 6 | 10 | 19
  Spain | 9 | 14 | 12 | 35

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved a Best Response of Complete Response, Partial Response, and Stable Disease (CR+PR+SD) (Clinical Benefit Rate)
Description: Clinical benefit rate is defined as the rate of confirmed CR, confirmed PR, and SD for 24 weeks duration and is the best response CR, PR, or SD as classified by the investigators according to the RECIST v1.1. CR is a disappearance of all target and non-target lesions and normalization of tumor marker level. PR is an at least 30% decrease in the sum of the diameters of target lesions (taking as reference the baseline sum diameter) without progression of not-target lesions or appearance of new lesions. SD is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease, taking as reference the smallest sum diameter since treatment started. Kaplan-Meier (KM) techniques were used to assess the time-to-event endpoints. Progressive Disease (PD) was defined as having at least 20% increase in sum of longest diameter of target lesions and minimum 5 mm increase above nadir.
Time Frame: Baseline to Measured Progressive Disease or Study Discontinuation (Up to 24 Weeks)
Population: All randomized participants who received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Enzastaurin + Fulvestrant QD + BID: Participants received Enzastaurin loading dose of 1125 mg, on Day 1 of Cycle 1 only then received Enzastaurin 500 mg orally (QD) once daily in a 28-day cycle.
  Participants received enzastaurin loading dose of 1125 mg, on Day 1 of Cycle 1 only then received Enzastaurin 250 mg orally (BID) twice daily in a 28-day cycle.
  Fulvestrant was given intramuscularly at a loading dose of 500 mg on Day 1 and 250 mg on Day 15 in Cycle 1. Subsequent doses of Fulvestrant 250 mg were given on Day 1 of Cycle 2 and every 28 days thereafter.
  .
- Enzastaurin + Fulvestrant BID: Participants received enzastaurin (250 mg; 2 tablets) or placebo administered orally twice daily (BID) in a 28-day cycle, until disease progression. Fulvestrant was given intramuscularly at a loading dose of 500 mg on Day 1 and 250 mg on Day 15 in Cycle 1. Subsequent doses of Fulvestrant 250 mg were given on Day 1 of Cycle 2 and every 28 days thereafter.
- Enzastaurin + Fulvestrant QD: Participants received Enzastaurin once daily (QD) regimen consisted of enzastaurin 500 mg orally QD in a 28-day cycle until disease progression. Fulvestrant was given intramuscularly at a loading dose of 500 mg on Day 1 and 250 mg on Day 15 in Cycle 1. Subsequent doses of Ful 250 mg were given on Day 1 of Cycle 2 and every 28 days thereafter.
Arm/Group | Enzastaurin + Fulvestrant QD + BID | Enzastaurin + Fulvestrant BID | Enzastaurin + Fulvestrant QD | Fulvestrant + Placebo
Number analyzed (Participants) | 94 | 39 | 55 | 58
percentage of participants | 43.6 [33.4 to 54.2] | 43.6 [27.8 to 60.4] | 43.6 [30.3 to 57.7] | 44.8 [31.7 to 58.5]
Statistical Analysis 1: Comparison: Enzastaurin + Fulvestrant QD + BID vs Fulvestrant + Placebo; Test type: Superiority; p = 0.6238, Fisher Exact
Statistical Analysis 2: Comparison: Enzastaurin + Fulvestrant BID vs Fulvestrant + Placebo; Test type: Superiority; p = 0.6282, Fisher Exact
Statistical Analysis 3: Comparison: Enzastaurin + Fulvestrant QD vs Fulvestrant + Placebo; Test type: Superiority; p = 0.6242, Fisher Exact

2. Secondary Outcome: Percentage of Participants Achieving Overall Tumor Response Complete Response (CR) or Partial Response (PR) [Overall Response Rate (ORR])
Description: The ORR is equal to the percentage of participants achieving a best overall response of partial response or complete response (PR + CR), according to RECIST version 1.1 criteria. CR was defined as the disappearance of all target and non-target lesions and any pathological lymph nodes must have reduction in short axis to <10 millimeter (mm) and normalization of tumor marker level of non-target lesions; PR was defined as having at least a 30% decrease in sum of longest diameter of target lesions; PD was defined as having at least 20% increase in sum of longest diameter of target lesions and minimum 5 mm increase above nadir; SD was defined as small changes that did not meet above criteria. Participants who had no post baseline tumor assessments were considered non-responders and included in the denominator when calculating response rate. The 95% confidence interval (CI) was calculated by exact method. Kaplan-Meier (KM) techniques were used to assess the time-to-event endpoints.
Time Frame: Baseline to Measured Progressive Disease or Study Discontinuation (Up to 24 Weeks)
Population: All randomized participants who received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Enzastaurin + Fulvestrant QD + BID | Enzastaurin + Fulvestrant BID | Enzastaurin + Fulvestrant QD | Fulvestrant + Placebo
Number analyzed (Participants) | 94 | 39 | 55 | 58
percentage of participants | 5.3 [1.7 to 12.0] | 5.1 [0.6 to 17.3] | 5.5 [1.1 to 15.1] | 5.2 [1.1 to 14.4]
Statistical Analysis 1: Comparison: Enzastaurin + Fulvestrant QD + BID vs Fulvestrant + Placebo; Test type: Superiority; p = 0.6390, Fisher Exact
Statistical Analysis 2: Comparison: Enzastaurin + Fulvestrant BID vs Fulvestrant + Placebo; Test type: Superiority; p = 0.6721, Fisher Exact
Statistical Analysis 3: Comparison: Enzastaurin + Fulvestrant QD vs Fulvestrant + Placebo; Test type: Superiority; p = 0.6349, Fisher Exact

3. Secondary Outcome: Duration of Clinical Benefit
Description: The duration of clinical benefit was measured from the time of clinical benefit of CR, PR or SD to the time of progressive disease or death from any cause. PD was defined as having at least 20% increase in sum of longest diameter of target lesions and minimum 5 mm increase above nadir. Kaplan-Meier (KM) techniques were used to assess the time-to-event endpoints.
Time Frame: Time of Clinical Benefit to Progressive Disease or Death (Up to 3 Years)
Population: All randomized participants who received at least one dose of study drug and had evaluable clinical benefit duration data.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Enzastaurin + Fulvestrant BID + QD: Participants received Enzastaurin loading dose of 1125 mg, on Day 1 of Cycle 1 only then received Enzastaurin 500 mg orally (QD) once daily in a 28-day cycle.
  Participants received enzastaurin loading dose of 1125 mg, on Day 1 of Cycle 1 only then received Enzastaurin 250 mg orally (BID) twice daily in a 28-day cycle.
  Fulvestrant was given intramuscularly at a loading dose of 500 mg on Day 1 and 250 mg on Day 15 in Cycle 1. Subsequent doses of Fulvestrant 250 mg were given on Day 1 of Cycle 2 and every 28 days thereafter.
  .
- Enzastaurin + Fulvestrant QD: Participants received Enzastaurin once daily (QD) regimen consisted of enzastaurin 500 mg orally QD in a 28-day cycle, until disease progression.
  Fulvestrant was given intramuscularly at a loading dose of 500 mg on Day 1 and 250 mg on Day 15 in Cycle 1. Subsequent doses of Ful 250 mg were given on Day 1 of Cycle 2 and every 28 days thereafter.
Arm/Group | Enzastaurin + Fulvestrant BID + QD | Enzastaurin + Fulvestrant BID | Enzastaurin + Fulvestrant QD | Placebo + Fulvestrant BID
Number analyzed (Participants) | 41 | 17 | 24 | 26
months | 9.6 [8.2 to 11.0] | 9.4 [7.4 to 12.2] | 9.6 [7.9 to 11.1] | 9.7 [7.4 to 12.6]
Statistical Analysis 1: Comparison: Enzastaurin + Fulvestrant BID + QD vs Placebo + Fulvestrant BID; Test type: Superiority; p = 0.8582, Log Rank
Statistical Analysis 2: Comparison: Enzastaurin + Fulvestrant BID vs Placebo + Fulvestrant BID; Test type: Superiority; p = 0.7307, Log Rank
Statistical Analysis 3: Comparison: Enzastaurin + Fulvestrant QD vs Placebo + Fulvestrant BID; Test type: Superiority; p = 0.9798, Log Rank

4. Secondary Outcome: Progression Free Survival (PFS)
Description: Progression-free survival (PFS) time was defined as the time from baseline to the first date of progressive disease (symptomatic or objective) or death due to any cause, whichever occurred first. PD was defined as having at least 20% increase in sum of longest diameter of target lesions and minimum 5 mm increase above nadir.For participants who were not known to have died or progressed as of the data-inclusion cutoff date, PFS time was censored at the date of the last objective progression-free disease assessment prior to the date of any subsequent systematic anticancer therapy. PFS was summarized using Kaplan-Meier estimates.
Time Frame: Baseline to Measured Progressive Disease or Death Due to Any Cause (Up to 3 Years)
Population: All randomized participants who had received at least one dose of study drug and had evaluable PFS data. Participants were censored in Fulvestrant + Enzastaurin (QD) arm = 4, the Fulvestrant + Enzastaurin (BID) arm = 6, and the Fulvestrant + Placebo arm = 6.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Enzastaurin + Fulvestrant QD + BID: Participants received Enzastaurin loading dose of 1125 mg, on Day 1 of Cycle 1 only then received Enzastaurin 500 mg orally (QD) once daily in a 28-day cycle.
  Participants received enzastaurin loading dose of 1125 mg, on Day 1 of Cycle 1 only then received Enzastaurin 250 mg orally (BID) twice daily in a 28-day cycle.
  Fulvestrant was given intramuscularly at a loading dose of 500 mg on Day 1 and 250 mg on Day 15 in Cycle 1. Subsequent doses of Fulvestrant 250 mg were given on Day 1 of Cycle 2 and every 28 days thereafter.
Arm/Group | Enzastaurin + Fulvestrant QD + BID | Enzastaurin + Fulvestrant BID | Enzastaurin + Fulvestrant QD | Fulvestrant + Placebo
Number analyzed (Participants) | 94 | 39 | 55 | 58
months | 5.2 [3.5 to 7.4] | 3.7 [2.8 to 7.4] | 6.0 [2.8 to 7.9] | 5.5 [3.8 to 7.4]
Statistical Analysis 1: Comparison: Enzastaurin + Fulvestrant QD + BID vs Fulvestrant + Placebo; Test type: Superiority; p = 0.5887, Log Rank
Statistical Analysis 2: Comparison: Enzastaurin + Fulvestrant BID vs Fulvestrant + Placebo; Test type: Superiority; p = 0.4516, Log Rank
Statistical Analysis 3: Comparison: Enzastaurin + Fulvestrant QD vs Fulvestrant + Placebo; Test type: Superiority; p = 0.7965, Log Rank

5. Secondary Outcome: Number of Participants Who Discontinued With Adverse Events (AE) and Serious Adverse Events (SAEs)
Description: Clinically significant events were defined as serious AEs (SAEs) and other non-serious AEs, regardless of causality. A summary of SAEs and other non-serious AEs, regardless of causality, is located in the Reported Adverse Events module. Participants who discontinued due to an AE or SAE are reported.
Time Frame: From Baseline to Study Completion (Up to 3 years, 9 months)
Population: All randomized participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Enzastaurin + Fulvestrant QD + BID | Enzastaurin + Fulvestrant BID | Enzastaurin + Fulvestrant QD | Fulvestrant + Placebo
Number analyzed (Participants) | 94 | 39 | 55 | 58
Participants
  Adverse Events (AEs) | 3 | 1 | 2 | 1
  Serious Adverse Events (SAEs) | 0 | 0 | 0 | 1

6. Secondary Outcome: Percentage of Participants With Enzastaurin Biomarkers and Disease State
Time Frame: Baseline, Cycle 2 to Study Completion (Up to 3 Years, 9 Months)
Population: Zero participants were analyzed due to insufficient samples being collected.
Arm/Group | Enzastaurin + Fulvestrant QD + BID | Enzastaurin + Fulvestrant BID | Enzastaurin + Fulvestrant QD | Fulvestrant + Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From Baseline to Study Completion (Up to 3 Years, 9 Months)
Description: All randomized participants who received at least one dose of study drug in Enzastaurin and Fulvestrant administered in combination or alone.
Groups:
- Fulvestrant + Enzastaurin (QD + BID): Participants received Enzastaurin loading dose of 1125 mg, on Day 1 of Cycle 1 only then received Enzastaurin 500 mg orally (QD) once daily in a 28-day cycle.
  Participants received enzastaurin loading dose of 1125 mg, on Day 1 of Cycle 1 only then received Enzastaurin 250 mg orally (BID) twice daily in a 28-day cycle.
  Fulvestrant was given intramuscularly at a loading dose of 500 mg on Day 1 and 250 mg on Day 15 in Cycle 1. Subsequent doses of Fulvestrant 250 mg were given on Day 1 of Cycle 2 and every 28 days thereafter.
- Fulvestrant + Enzastuarin (QD): Participants received enzastaurin (250 mg; 2 tablets) or placebo administered orally twice daily (BID) in a 28-day cycle, until disease progression. Fulvestrant was given intramuscularly at a loading dose of 500 mg on Day 1 and 250 mg on Day 15 in Cycle 1. Subsequent doses of Fulvestrant 250 mg were given on Day 1 of Cycle 2 and every 28 days thereafter.
- Fulvestrant + Enzastuarin (BID): Participants received Enzastaurin once daily (QD) regimen consisted of enzastaurin 500 mg orally QD in a 28-day cycle until disease progression. Fulvestrant was given intramuscularly at a loading dose of 500 mg on Day 1 and 250 mg on Day 15 in Cycle 1. Subsequent doses of Ful 250 mg were given on Day 1 of Cycle 2 and every 28 days thereafter.
Arm/Group | Fulvestrant + Enzastaurin (QD + BID) | Fulvestrant + Enzastuarin (QD) | Fulvestrant + Enzastuarin (BID) | Fulvestrant + Placebo
Serious Adverse Events (participants affected / at risk) | 17/94 | 9/39 | 8/55 | 11/58
Other Adverse Events (participants affected / at risk) | 78/94 | 31/39 | 47/55 | 50/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fulvestrant + Enzastaurin (QD + BID) (N=94) | Fulvestrant + Enzastuarin (QD) (N=39) | Fulvestrant + Enzastuarin (BID) (N=55) | Fulvestrant + Placebo (N=58)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ischaemic cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Asthenia (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Disease progression (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Metastases to skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ureteric dilatation (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Phlebitis (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fulvestrant + Enzastaurin (QD + BID) (N=94) | Fulvestrant + Enzastuarin (QD) (N=39) | Fulvestrant + Enzastuarin (BID) (N=55) | Fulvestrant + Placebo (N=58)
Anaemia (Blood and lymphatic system disorders) | 8 (9) | 3 (3) | 5 (6) | 4 (4)
Vertigo (Ear and labyrinth disorders) | 2 (3) | 0 (0) | 2 (3) | 4 (4)
Abdominal pain (Gastrointestinal disorders) | 8 (11) | 3 (5) | 5 (6) | 4 (4)
Abdominal pain upper (Gastrointestinal disorders) | 7 (9) | 3 (3) | 4 (6) | 2 (2)
Constipation (Gastrointestinal disorders) | 17 (21) | 7 (10) | 10 (11) | 7 (9)
Diarrhoea (Gastrointestinal disorders) | 20 (33) | 6 (16) | 14 (17) | 10 (12)
Dry mouth (Gastrointestinal disorders) | 3 (3) | 2 (2) | 1 (1) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 4 (4) | 3 (3) | 1 (1) | 2 (2)
Faeces discoloured (Gastrointestinal disorders) | 3 (3) | 2 (2) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Nausea (Gastrointestinal disorders) | 31 (33) | 13 (13) | 18 (20) | 18 (31)
Vomiting (Gastrointestinal disorders) | 9 (10) | 4 (4) | 5 (6) | 6 (8)
Asthenia (General disorders) | 15 (19) | 6 (9) | 9 (10) | 10 (11)
Chest pain (General disorders) | 3 (4) | 0 (0) | 3 (4) | 5 (5)
Fatigue (General disorders) | 21 (23) | 9 (9) | 12 (14) | 11 (14)
Influenza like illness (General disorders) | 4 (4) | 2 (2) | 2 (2) | 1 (1)
Malaise (General disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 6 (7) | 3 (4) | 3 (3) | 3 (3)
Pyrexia (General disorders) | 7 (8) | 4 (5) | 3 (3) | 3 (3)
Bronchitis (Infections and infestations) | 4 (8) | 2 (5) | 2 (3) | 4 (4)
Cystitis (Infections and infestations) | 5 (5) | 3 (3) | 2 (2) | 2 (2)
Infection (Infections and infestations) | 4 (5) | 2 (3) | 2 (2) | 2 (2)
Nasopharyngitis (Infections and infestations) | 5 (5) | 0 (0) | 5 (5) | 0 (0)
Pharyngitis (Infections and infestations) | 2 (3) | 2 (3) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 3 (3) | 0 (0) | 3 (3) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 4 (5)
Alanine aminotransferase increased (Investigations) | 4 (4) | 1 (1) | 3 (3) | 0 (0)
Electrocardiogram qt prolonged (Investigations) | 3 (5) | 0 (0) | 3 (5) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 4 (4) | 1 (1) | 3 (3) | 1 (1)
Weight decreased (Investigations) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 5 (5) | 2 (2) | 3 (3) | 2 (2)
Hypercalcaemia (Metabolism and nutrition disorders) | 3 (3) | 3 (3) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 (10) | 7 (7) | 2 (3) | 7 (8)
Back pain (Musculoskeletal and connective tissue disorders) | 8 (8) | 5 (5) | 3 (3) | 7 (7)
Bone pain (Musculoskeletal and connective tissue disorders) | 9 (9) | 2 (2) | 7 (7) | 10 (11)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 3 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 2 (2) | 5 (5)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (5) | 0 (0) | 5 (5) | 2 (2)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 2 (2) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 3 (5) | 3 (5) | 0 (0) | 5 (5)
Headache (Nervous system disorders) | 11 (14) | 4 (5) | 7 (9) | 7 (8)
Paraesthesia (Nervous system disorders) | 3 (4) | 2 (3) | 1 (1) | 1 (1)
Sciatica (Nervous system disorders) | 3 (3) | 0 (0) | 3 (3) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (2) | 1 (1) | 1 (1) | 3 (4)
Chromaturia (Renal and urinary disorders) | 9 (9) | 3 (3) | 6 (6) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 2 (2) | 7 (7) | 7 (8)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1) | 3 (3) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 12 (14) | 4 (5) | 8 (9) | 8 (8)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 2 (2) | 4 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (4) | 3 (3) | 1 (1) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (1) | 3 (3) | 3 (3)
Hot flush (Vascular disorders) | 14 (17) | 8 (9) | 6 (8) | 5 (7)

LIMITATIONS AND CAVEATS:
The translational research component of the study was cancelled due to lack of efficacy in the experimental arm. Due to an amendment to the initial therapy, 250 mg BID dosing was added to the design of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days